CLINICAL TRIAL: NCT05887791
Title: Clinical Study to Assess the Effect of a Collagen Hydrolysate on Postprandial Blood Glucose Profile in Prediabetic and Healthy Subjects: Randomized, Double-blind, Placebo-controlled, Cross-over Study With Different Dosages
Brief Title: Effect of a Collagen Hydrolysate on Postprandial Blood Glucose Profile in Prediabetic and Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rousselot BVBA (Industry)
Collaborators: BioTeSys GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: BTS1984/23
Record Dates: First submitted 2023-05-24; First posted 2023-06-05 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2023-06

CONDITIONS: Healthy; Prediabetic State
Keywords: collagen peptides; blood sugar modifying
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Collagen hydrolysate dose 1 (Experimental): Source: porcine; standardized to 10 g provided as single dose. Orally applied in flavoured water.
  Interventions: Dietary Supplement: Collagen hydrolysate
- Collagen hydrolysate dose 2 (Experimental): Source: porcine; standardized to 5 g provided as single dose. Orally applied in flavoured water.
  Interventions: Dietary Supplement: Collagen hydrolysate
- Placebo (Placebo Comparator): Flavoured water
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Collagen hydrolysate — Single dose
  Arms: Collagen hydrolysate dose 1; Collagen hydrolysate dose 2
Other: Placebo — Single dose
  Arms: Placebo

SUMMARY:
To investigate the effect of two different dosages collagen hydrolysate (CH) on postprandial blood glucose and insulin profile in prediabetic and normo-glycaemic subjects.This will be investigated in a cross-over randomized double-blind placebo controlled study design.

ELIGIBILITY:
Main Inclusion Criteria:

* Prediabetic subjects: Male and female subjects with prediabetic HbA1c values between 5.7% and 6.4% and/or fasting glucose ≥ 100 mg/dL and ≤ 125 mg/dL (in venous plasma) (twice confirmed at two independent days if HbA1c is < 5.7%) or Healthy normo-glycaemic subjects: fasting glucose <100 mg/dL and HbA1c is < 5.7%
* Age: 18-70 years
* Body mass index 19-35 kg/m2
* Current Non-smoker
* Signed informed consent form
* No changes in food habits or physical activity 3 months prior to screening and during the study
* If applicable, stable intake of chronic medication of at least 4 weeks

Main Exclusion Criteria:

* Subjects with diagnosed Type 2 Diabetes mellitus with medical treatment
* Presence of disease or drug(s) influencing digestion (incl. recent intake of antibiotics) and absorption of nutrients
* Intake of medications known to affect glucose tolerance, e.g., diabetic medication, SGLT-2 inhibitors, GLP-1 receptor agonists, steroids, protease inhibitors or antipsychotics
* Chronic intake of substances affecting blood coagulation (e.g. acetylic acid (100 mg as standard prophylactic treatment allowed when dose is stable 1 month prior to screening), anticoagulants, diuretics, thiazides (diuretics and thiazides allowed e.g. for hypertension treatment when dose is stable 1 month prior to screening)), which in the Investigator's opinion would impact patient safety
* Severe liver or renal disease or laboratory evidence of hepatic dysfunction (i.e. alkaline phosphatase, ALT, AST >3 x ULN)
* Known inflammatory or malignant gastrointestinal diseases (i.e. colitis ulcerosa, Morbus Crohn, celiac disease, malignant diseases e.g. colon-cancer, rectum cancer, pancreatitis)
* Clinically relevant findings as established by medical history, physical examination, clinical laboratory and/or vital signs
* Intake of food supplements known to affect glucose tolerance, e.g., cinnamon capsules, conjugated linoleic acids
* Drug-, alcohol- and medication abuses
* Pregnant or breast-feeding women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-12-23 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Glucose iAUC | 0-180 minutes postprandially
  Area under the curve (AUC) calculated as the incremental area under the blood glucose response curve, ignoring the area beneath the fasting concentration: Glucose-iAUC(0-180minutes)

SECONDARY OUTCOMES:
Glucose iAUC | 0-240 minutes postprandially
  Area under the curve calculated as the incremental area under the blood glucose response curve, ignoring the area beneath the fasting concentration: Glucose-iAUC(0-240minutes)
Glucose Cmax | 0-180 minutes postprandially
  Maximum blood glucose concentration (Cmax)
Delta Cmax | 0-180 minutes postprandially
  Maximum increase of blood glucose concentration
Tmax | 0-180 minutes postprandially
  Time to reach maximum blood glucose concentration (Tmax)
T baseline | 0-240 minutes postprandially
  First time to reach baseline again after increase or decrease in blood glucose
Matsuda-Index | 0-120 minutes postprandially
  Determination of Insulin sensitivity
Glucose dip | 0-240 minutes postprandially
  maximum dip below baseline and time point of glucose dip
Insulin iAUC | up to 0-240 minutes postprandially
  Area under the curve calculated as the incremental area under the insulin curve
GLP-1 | 0-120 minutes postprandially
  Incretin response (Glucagon-like Peptide-1)
Satiety assessment | 0-240 minutes postprandially
  Visual analog scale (VAS) Scale (0: not at all 100: extremely)

OTHER OUTCOMES:
Gastrointestinal hormones | 0-120 minutes postprandially
  Peptid YY (PYY), Ghrelin, Cholecystokinin (CCK), Leptin
Amino acids | 0-240 minutes postprandially
  Concentration-time curve of amino acids in plasma together with small molecular weight peptides

CONTACTS AND LOCATIONS:
Overall Officials: Nicoletta Virgilio, PhD, Study Director — Rousselot BV
Locations (1):
- BioTeSys GmbH, Esslingen am Neckar, Germany

IPD SHARING:
Plan to Share IPD: No